CLINICAL TRIAL: NCT01304290
Title: Glucose/Insulin Clamp on Solid Organ Transplant (Liver, Kidney, Pancreas and Heart) on Cadaveric Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, peter metrakos, Director Multiorgan Transplant Program-MUHC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SDR-09-054
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Complication of Transplanted Organ, Nos
Keywords: inflammatory process; hyperglycaemia; inflammatory cytokine response; organ survival; hyperinsulinemic clamp
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention)
- Glucose/Insulin Clamp (Experimental)
  Interventions: Other: Hyperinsulinemic/normoglycemic clamp

INTERVENTIONS:
Other: Hyperinsulinemic/normoglycemic clamp — Dextrose/insulin therapy will start. Dextrose and insulin are given using the so-called "normoglycemic, hyperinsulinemic clamp". Plasma insulin concentration will be increased by a 2ìU/kg/min continuous infusion of insulin. Dextrose will be infused at the rate required to maintain normoglycemia (4-6 mmol/l) until cross clamping of the aorta. The dextrose/insulin therapy will be maintained for a time period of minimum 6 hours.
  Other Names: no brand name; its dextrose D20%
  Arms: Glucose/Insulin Clamp

SUMMARY:
Our objective in this study will be to determine if implementing the glucose/insulin clamp (GICT) on cadaveric organ donors can:

* Prevent hyperglycaemia
* Drop in the inflammatory cytokine response after brain death after a minimum of 6 hours therapy with the GICT prior to organ procurement.
* Assess organ (heart, liver, pancreas and kidney) survival at one year post-transplant
* Assess graft function by evaluating:

  * Liver: post-transplant liver function score (PTLF)
  * Kidney: graft function as defined by UNOS (immediate graft function IGF, slow graft function SGF and delayed graft function DGF and
  * Pancreas: 7 day post-transplant insulin requirement, C-peptide and C-RP levels at day one and seven post-transplantation

ELIGIBILITY:
Inclusion Criteria:

* Donors must be over 18 years of age
* Brain death donors only
* Getting consent prior to any specific protocol procedure under Transplant Quebec regulations.

Exclusion Criteria:

* Inability to obtain a research consent
* Time interval between the start of the study and cross-clamping less than 6 hours.
* No solid organs retrieved for transplantation
* Diagnosed with Type 1 Diabetes
* Donor has uncontrolled serum blood glucose levels (above 10 mmol/L) at time of inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
• Drop in the inflammatory cytokine response after brain death after a minimum of 6 hours therapy with the GICT prior to organ procurement. | during transplant
  Our objective in this study will be to determine if implementing the glucose/insulin clamp (GICT) on cadaveric organ donors can:
  * Prevent hyperglycaemia
  * Drop in the inflammatory cytokine response after brain death after a minimum of 6 hours therapy with the GICT prior to organ procurement.

SECONDARY OUTCOMES:
Assess organ (heart, liver, pancreas and kidney) survival at one year post-transplant | 1 year post-transplant
  * Assess organ (heart, liver, pancreas and kidney) survival at one year post-transplant
  * Assess graft function by evaluating:
    * Liver: post-transplant liver function score (PTLF)
    * Kidney: graft function as defined by UNOS (immediate graft function IGF, slow graft function SGF and delayed graft function DGF and
    * Pancreas: 7 day post-transplant insulin requirement, C-peptide and C-RP levels at day one and seven post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Peter Metrakos, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada